CLINICAL TRIAL: NCT01124357
Title: A Randomised Control Trial To Compare the Effectiveness of Outpatient Endometrial Ablation Techniques (Novasure vs Thermachoice)in the Treatment of Menorhagia
Brief Title: A Study to Compare the Effectiveness of Two Different Outpatient Endometrial Ablation Techniques Used for Heavy Periods
Acronym: COAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Mr Justin Clark, Birmingham Women's NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLA004.
Record Dates: First submitted 2010-03-18; First posted 2010-05-17 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2006-05

CONDITIONS: Menorrhagia
Keywords: Heavy menstrual bleeding; menorrhagia; ThermachoiceTM; NovaSureTM; Endometrail Ablation
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- novasure (Active Comparator): Bipolar radio-frequency energy ablation of the endometrium by thermal therapy under impedance control. The bipolar current generated by the device produces a tapered depth of ablation with shallower ablation in the cornual regions / lower uterine segment and a deeper ablation in the mid-body of the uterus..
  Interventions: Device: NovaSure
- thermachoice (Other): ThermachoiceTM III thermal balloon ablation
  Interventions: Device: thermachoice

INTERVENTIONS:
Device: NovaSure — Bipolar radio-frequency energy ablation of the endometrium by thermal therapy under impedance control. The bipolar current generated by the device produces a tapered depth of ablation with shallower ablation in the cornual regions / lower uterine segment and a deeper ablation in the mid-body of the uterus..
  Other Names: Bipolar radio-frequency energy ablation
  Arms: novasure
Device: thermachoice — ThermachoiceTM III thermal balloon ablation
  Other Names: Thermal balloon ablation
  Arms: thermachoice

SUMMARY:
STUDY HYPOTHESIS: Does outpatient NovaSureTM endometrial ablation alleviate excessive menstrual bleeding and improve life quality more effectively than outpatient ThermachoiceTM endometrial ablation?

DETAILED DESCRIPTION:
Heavy menstrual bleeding (HMB) or 'menorrhagia' is a common condition with a major impact on health-related quality of life and health resource utilization in both primary and secondary care. In over 50% of cases no organic pathology is present and the term dysfunctional uterine bleeding (DUB) is used. First line treatment of DUB is medical and where this fails, surgery is indicated using either minimally invasive approaches (endometrial ablation) or major surgery (hysterectomy). Endometrial ablation has been extensively evaluated against the gold standard of hysterectomy and shown to be effective and associated with fewer complications. The technique involves destroying the entire, or a substantial proportion, of the endometrium thereby preventing cyclical endometrial regeneration and suppressing or reducing menstrual blood loss. Recent advances in endoscopic technology have resulted in the development of miniature, automated ablative systems (so called 'second generation devices'), which are easy to use, safe and obviate the need for routine unpleasant and expensive endometrial preparatory drugs10. Moreover, these devices have the potential to be routinely used in the outpatient or 'office' setting without the need for general anaesthesia. This approach is increasingly being advocated as it expands patient choice and potentially increasing safety and cost-effectiveness of treatment.

The three most commonly employed and evaluated ablative devices are ThermachoiceTM III thermal balloon ablation (Gynecare Inc, Somerville, NJ, USA), Microwave endometrial ablation (Microsulis plc, Waterlooville, Hampshire, UK) and NovaSureTM impedance-controlled endometrial ablation (Cytyc, Marlborough, MA USA). All appear to have comparable efficacy when employed as an inpatient under general anaesthesia in terms of patient satisfaction and life quality although data on direct head to head comparisons of these procedures when performed in an outpatient environment are scarce. All techniques have been employed without the need for general anaesthesia11,16-19, but only ThermachoiceTM has been reported in an outpatient setting11, without the need for formal theatre facilities or conscious sedation. The Microwave technique necessitates significant dilatation of the cervix that limits its potential for use in an outpatient setting in contrast to ThermachoiceTM and NovaSureTM10.

The newer NovasureTM system is more effective than ThermachoiceTM because inpatient studies report a higher rate of amenorrhoea (cessation of menstrual periods - 43% versus 8%). Moreover, NovaSureTM may be a better technique for use in conscious patients in an outpatient setting as it is a shorter procedure (1.5 versus 8 minutes) and associated with less post-operative pain16,19 but it does require a greater degree of potentially painful cervical dilatation10. There is thus a need for a randomised trial to compare the effectiveness and acceptability of ThermachoiceTM and NovaSureTM endometrial ablation in an outpatient setting for the treatment of menorrhagia.

ELIGIBILITY:
Inclusion Criteria:

* Women with no desire to preserve their fertility who have heavy menstrual bleeding without organic pathology (DUB) of more than six months duration
* Premenopausal follicular follicle stimulating hormone (FSH) level of less than 40 IU/L.
* Associated functional disability (negative impact on life quality).
* Lack of response to medical treatment.
* Prepared to undergo surgical treatment without general anaesthesia

Exclusion Criteria:

* Women under 25 years
* Suspected genital tract infection
* Uterine pathology including endometrial pathology on endometrial biopsy (e.g. endometrial hyperplasia or carcinoma) and structural lesions (e.g. uterine malformations, adhesions, polyps, submucous fibroids or extracavity fibroids > 3cm in diameter) as identified on pelvic ultrasound and/or outpatient hysteroscopy.
* Uterine cavity length >11cm
* Adnexal pathology
* Previous open myomectomy or endometrial ablation / resection and classical caesarian section
* patients considered vulnerable (e.g. current mental illness, emotionally labile, learning difficulties, immaturity)

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-05; Primary Completion 2007-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Amenorrhoea | 6 months after the intervention.
  The objective of any treatment for HMB is to substantially reduce the amount of menstrual blood loss.Amenorrhoea rates are often chosen as the primary outcome measure in clinical trial of the effectiveness of endometrial ablation in women with HMB.

SECONDARY OUTCOMES:
Visual analogue scale for assessment of pain | 24 hours
  The main limitation of outpatient interventions is the amount of pain generated. Endometrial ablation has been shown to be feasible and generally well tolerated in conscious patients in small observational series10-11, but direct randomised comparisons between techniques regarding the amount of pain experienced during surgery are lacking

CONTACTS AND LOCATIONS:
Overall Officials: Justin Mr Clark, MD MRCOG, Principal Investigator — Birmingham Women's NHS Foundation Trust

REFERENCES:
- [Derived] Smith PP, Malick S, Clark TJ. Bipolar radiofrequency compared with thermal balloon ablation in the office: a randomized controlled trial. Obstet Gynecol. 2014 Aug;124(2 Pt 1):219-225. doi: 10.1097/AOG.0000000000000395. PMID 25004347
- [Derived] Clark TJ, Samuel N, Malick S, Middleton LJ, Daniels J, Gupta JK. Bipolar radiofrequency compared with thermal balloon endometrial ablation in the office: a randomized controlled trial. Obstet Gynecol. 2011 Jan;117(1):109-118. doi: 10.1097/AOG.0b013e3182020401. PMID 21173651